CLINICAL TRIAL: NCT02874313
Title: Effect of Continuous Positive Airway Pressure on the Progression of Vascular Retinal Disease in Patients With Sleep Apnea and Non-proliferative Diabetic Retinopathy. A Randomized Clinical Trial
Brief Title: CPAP Effect on the Progression of Diabetic Retinopathy in Patients With Sleep Apnea
Acronym: RetinAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Francisco Garcia-Rio, MD, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HULP PI-2476
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Diabetic Retinopathy; Sleep Apnea
Keywords: CPAP; Sleep apnea; Diabetes; Diabetic retinopathy
MeSH Terms: conditions — Diabetic Retinopathy; Sleep Apnea Syndromes; Diabetes Mellitus | interventions — Continuous Positive Airway Pressure; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP treatment (Experimental): Diet and conventional pharmacological treatment with oral antidiabetic drugs or insulin plus continuous positive airway pressure (CPAP)
  Interventions: Device: Continuous positive airway pressure; Drug: Pharmacological treatment; Other: Conventional anti-diabetic diet recommendations
- Control treatment (Active Comparator): Diet and conventional pharmacological treatment with oral antidiabetic drugs or insulin
  Interventions: Drug: Pharmacological treatment; Other: Conventional anti-diabetic diet recommendations

INTERVENTIONS:
Device: Continuous positive airway pressure — Nocturnal continuous positive airway pressure by a nasal mask. CPAP pressure will be automatically titrated using a AutoSet device (ResMed).
  Arms: CPAP treatment
Drug: Pharmacological treatment — Conventional pharmacological treatment with oral antidiabetic drugs or insulin
Other: Conventional anti-diabetic diet recommendations

SUMMARY:
Objectives: Main objective: To compare the percentage of patients with new microaneurysm or hard exudates after 12 months between the CPAP group and the control group. Secondary objectives: To compare the central macula volume, ganglion cell layer thickness and central fovea thickness at baseline and 12, 24 and 52 weeks after randomization between the two study groups; to compare the percentage of patients who have an improvement loss of visual acuity (more than or equal to 15 letters in patients with macular edema and more than or equal to five letters in patients without macular edema) among the baseline visit and the weeks 12, 24 and 52 between the two study groups; to compare the percentage of patients who reach a higher level of diabetic retinopathy at 54 weeks between the two study groups; to compare the resolution time of central macula thickness from the randomization between the two study groups; to compare the glycated hemoglobin at baseline and 12, 24 and 52 weeks after randomization between the two study groups; and to compare the serum levels of inflammatory cytokines, oxidative stress biomarkers, sympathetic tone, and intake regulator hormones at baseline and 12 and 52 weeks after randomization between the two study groups.

Methodology: Randomized, multicenter, non-blinded, parallel groups, conventional treatment-controlled trial of 12 months of duration.

Subjects will randomize to conventional dietary and pharmacological treatment or conventional dietary and pharmacological treatment plus continuous positive airway pressure (CPAP). Study subjects: Subjects 35 to 75 years with type 2 diabetes and a clinical diagnosis of mild diabetic retinopathy (with or without macular edema), better visual acuity from 20/40 to 20/320 letters and refraction with a spherical equivalent less than ± 5 diopter.

Efficacy variables: Thickness of the central sub-field, central subfield volume, ganglion cell layer thickness, and presence of clinical or subclinical macular edema, serous retinal or retinal pigment epithelium detachment, intraretinal cysts or haemorrhages assessed by optical coherence tomography; presence of cotton exudates, microhemorrhages, microaneurysms, , microvascular retinal abnormalities, or a vein/artery ratio > 2/1 in examination of ocular fundus/retinography; better corrected visual acuity; glycosylated hemoglobin (HbA1c); fasting glucose and insulin; homeostatic model assessment (HOMA) and QUICKI indices; lipid profile, troponin I, proBNP, homocysteine and C-reactive protein; systemic biomarkers of inflammation, oxidative stress, endothelial damage, sympathetic activity and appetite-regulating hormones and clinical questionnaires: short form (SF)-12, visual function questionnaire (VFQ25) and iPAQ.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 35 to 75 years old.
* Previous diagnosis of type 2 diabetes, fulfilling at least one of the following criteria: 1) current treatment with oral antidiabetic drugs and/or insulin; 2) a fasting glucose value above 126 mg/dl on at least 2 occasions; 3) blood glucose level at 2 hours after an oral glucose tolerance test is equal to or more than 200 mg/dl; or 4) a glycated hemoglobin (HbA1c) level > 6.5 %
* Clinical diagnosis of mild non-proliferative diabetic retinopathy, with or without macular edema.
* Best corrected visual acuity according to ETDRS optotype from 20/40 to 20/320 letters from 4 meters (score 73-25 letters) in the studied eye.
* Spherical equivalent refraction less than ± 5 dioptre.

Exclusion Criteria:

* Prior systemic treatment for diabetic retinopathy, with the exception of nutritional supplements or vitamins.
* Pre-treatment with anti-vascular endothelial growth factor (VEGF) drugs in the studied eye. It is allowed a pre-treatment with anti-VEGF approved in the other eye more than 3 months ago.
* Prior systemic anti-VEGF, experimental or approved treatment, three months before the inclusion.
* Evidence of inflammation or infection in or around the studied eye.
* Treatment with troglitazone in the last three months.
* Eye surgery (including cataract surgery) in the studied eye three months before the inclusion.
* Late macular degeneration (geographical with foveal or neovascular involvement).
* Vascular retinal diseases, such as vascular occlusions.
* Previous diagnosis of other eye diseases that could lead to a decrease in visual acuity.
* Systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mm Hg at the baseline visit.
* Stroke, transient ischemic attack, acute coronary syndrome, or hospitalization for heart failure worsening, within the previous 30 days.
* Professional drivers, risk profession or respiratory failure.
* Severe daytime sleepiness (Epworth sleepiness scale >18)
* Concomitant treatment with high doses of acetylsalicylic acid (> 500 mg/day) or continuous treatment with non-steroidal anti-inflammatory drugs
* Previous treatment with CPAP
* Participation in another clinical trial within the 30 days prior to randomization.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-08; Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in of retinal microaneurysm or hard exudates | 12 months
  To compare the change in percentage of retinal microaneurysm or hard exudates between the patients allocated to CPAP group and the control group

SECONDARY OUTCOMES:
Change from baseline of the central macula volume | 3, 6 and 12 months
  To compare the change in central macula volume assessed by optical coherence tomography between the patients allocated to CPAP group and the control group
Change from baseline of the ganglion cell layer thickness | 3, 6 and 12 months
  To compare the change in ganglion cell layer thickness assessed by optical coherence tomography between the patients allocated to CPAP group and the control group
Change from baseline of the central fovea thickness | 3, 6 and 12 months
  To compare the change in the central fovea thickness assessed by optical coherence tomography between the patients allocated to CPAP group and the control group
Change from baseline of the severity level of diabetic retinopathy | 3, 6 and 12 months
  To compare the change in the severity level of diabetic retinopathy between the patients allocated to CPAP group and the control group
Change from baseline of the visual acuity | 12 months
  To compare the change in the visual acuity between the patients allocated to CPAP group and the control group
Change from baseline in glycated hemoglobin levels | 3, 6 and 12 months
  To compare the change in glycated hemoglobin levels between the patients allocated to CPAP group and the control group
Change form baseline in HOMA index | 3, 6 and 12 months
  To compare the change in HOMA index between the patients allocated to CPAP group and the control group
Change form baseline in QUICKI index | 3, 6 and 12 months
  To compare the change in QUICKI index between the patients allocated to CPAP group and the control group
Change from baseline in the health-related quality of life assessed by the VFQ25 questionnaire | 12 months
  To compare the change in the total score and the domains of the questionnaire VFQ25 between the CPAP group and the control group
Change from baseline in the health-related quality of life assessed by the SF-12 questionnaire | 12 months
  To compare the change in the total score and the domains of the questionnaire SF-12 between the CPAP group and the control group
Change from baseline in the daily physical activity of patients with diabetic retinopathy and obstructive sleep apnea | 12 months
  To compare the change in the total score of the International Physical Activity Questionnaire (iPAQ) between the CPAP group and the control group
Change form baseline in the plasmatic levels of biomarkers of inflammation | 12 months
  To compare the change in the plasmatic levels of interleukin (IL)-1beta, IL-6, IL-8 and tumor necrosis factor-alpha between the CPAP group and the control group
Change form baseline in the plasmatic levels of appetite-regulating hormones | 12 months
  To compare the change in the plasmatic levels of leptin and adiponectin between the CPAP group and the control group
Change form baseline in the plasmatic levels of endothelin | 12 months
  To compare the change in the plasmatic levels of endothelin, intercellular adhesion molecule-1 (ICAM-1) and vascular cell adhesion molecule-1 (VCAM-1) between the CPAP group and the control group
Change from baseline of intraocular pressure | 3, 6 and 12 months
  To compare the change in the intraocular pressure between the patients allocated to CPAP group and the control group

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Garcia-Rio, MD, Study Chair — Hospital Universitario La Paz, IdiPAZ
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia-Sanchez A, Villalain-Rodes I, Jaureguizar A, Zamarron E, Martinez-Ceron E, Casitas R, Galera R, Cubillos-Zapata C, Garcia J, Asencio M, Garcia-Rio F. Continuous Positive Airway Pressure Effect on Progression of Retinal Disease in Patients with Sleep Apnea and Nonproliferative Diabetic Retinopathy: A Randomized Clinical Trial. Ann Am Thorac Soc. 2024 Jan;21(1):102-113. doi: 10.1513/AnnalsATS.202304-296OC. PMID 37793101